CLINICAL TRIAL: NCT05404477
Title: Randomized Study of TransAeris® System for Enhanced Recovery After Surgery (ERAS) in Cardiac Surgery Patients in France at Risk of Prolonged Mechanical Ventilation
Brief Title: Study of TransAeris® System for Enhanced Recovery After Surgery in France
Acronym: ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 20-1000-108
Record Dates: First submitted 2022-05-13; First posted 2022-06-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Ventilator-Induced Diaphragm Dysfunction

STUDY DESIGN:
Intervention Model Description: This study is an open label, randomized, cross-over study in adult open cardiac surgery patients. All subjects will receive TransLoc electrodes at the time of open sternotomy cardiac procedure. Half of subjects will have TransAeris turned on upon entry to ICU, the other half will receive standard of care with TransAeris turned on if still intubated on mechanical ventilation after 120 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Other): Treatment with TransAeris stimulation upon completion of procedure
  Interventions: Device: TransAeris System
- Control (Other): Control subject will cross-over to treatment with the TransAeris System if still on mechanical ventilation at 120 hours post-op
  Interventions: Device: TransAeris System

INTERVENTIONS:
Device: TransAeris System — The TransAeris System includes four TransLoc® intramuscular diaphragm electrodes, the TransAeris external stimulator, and the FrictionLoc® connectors which provide the interface between the TransLoc electrodes and the TransAeris stimulator.

SUMMARY:
This study will be conducted as a randomized trial of the TransAeris system for the prevention and treatment of ventilator-induced diaphragm dysfunction (VIDD) in patients identified prior to surgery to be at greater risk of prolonged mechanical ventilation (PMV).

DETAILED DESCRIPTION:
This study is a monocentric and open label randomized study in adult open cardiac surgery patients. Eligible patients from whom informed consent is obtained are enrolled in the study. All subjects will be implanted with the TransLoc electrodes during their primary surgery. Patients are randomized to treatment or control groups prior to surgical placement of the TransLoc electrodes.

Comparison will be made between treatment and control patients during the initial 120 hours of study, then comparison of cross-over control patients' EMG from baseline to treatment.

Further comparison of MV Time, ventilator free days and other outcome measures will be made for all patients, over the course of the 30-day treatment period, to literature on an observational basis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing an open cardiac procedure by median sternotomy
2. Subject is at risk of prolonged mechanical ventilation according to one or more of the following criteria:

   1. Prior open cardiac surgery
   2. Left Ventricular Ejection Fraction (LVEF) ≤ 30%
   3. History of TIA or CVA
   4. Pre-operative or anticipated intraoperative intra-aortic balloon pump
   5. History of COPD
3. Subject is at least 22 years of age
4. Informed consent has been obtained from the subject
5. Subject is covered by a healthcare insurance

Exclusion Criteria:

1. Subject is on invasive mechanical ventilation prior to procedure
2. Subject has known or pre-existing phrenic nerve paralysis
3. Subject is having a left ventricular assist device (LVAD) implanted
4. Subject has progressive, non-reversible neuromuscular disease affecting the diaphragm
5. Subject is pregnant or lactating
6. Subject is actively participating in another clinical study which could affect outcomes in this study
7. Subject deprived of liberty
8. Subject under court protection

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Serious device-related adverse events | 60 days after implantation
  Number of serious device-related adverse effects
Time on mechanical ventilation | 90 days after study completion
  Time measured in hours on Mechanical Ventilation and Proportion of patients weaned at 48- and 120-hours post-op

SECONDARY OUTCOMES:
ICU Care | 90 days after study completion
  Number of instances of interference with ICU care
Device related adverse events | 90 days after study completion
  Number of Device related adverse events
Mortality | 90 days after study completion
  Mortality at 30-day post removal of electrodes
Mechanical ventilation time | 90 days after study completion
  Time on mechanical ventilation measured in hours from entry to the ICU and reversed paralytics
EMG | 90 days after study completion
  EMG analysis of cross-over patients
Ventilator Free Days | 90 days after study completion
  Number of days alive and free from mechanical ventilation
Length of stay | 90 days after study completion
  Number of days in the ICU and in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Henri David, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU - Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] David CH, Vourc'h M, Guimbretiere G, Mugniot A, Lacoste P, Cadiet J, Rozec B, Arora R, Pelletier M, Sabik J, Onders R. Multicentre Study of Diaphragm Pacing in High-Risk Cardiac Surgery to Decrease Postoperative Mechanical Ventilation. Eur J Cardiothorac Surg. 2026 Jan 6;68(1):ezaf472. doi: 10.1093/ejcts/ezaf472. PMID 41416899

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT05404477/Prot_SAP_000.pdf